CLINICAL TRIAL: NCT06349876
Title: Cholecystectomy in Patients With Silent Common Bile Duct Stones
Status: Completed | Type: Observational
Sponsor: Suez University (Other)
Responsible Party: Principal Investigator, Ahmad Ali Maklad, lecturer, Suez University
Other Study IDs: SUEZ MED - IRB Approval NO: 6
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Performing Cholecystectomy in Patients With Chronic Calcular Choleycystits
Keywords: CBD stones ,; cholecystectomy; silent stones
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lap chole: patients presented by cholecystitis with silent CBD stones
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — slandered laparoscopic cholecystectomy

SUMMARY:
Aim of this study is to evaluate the efficacy of performing only cholecystectomy in patients with asymptomatic common bile duct stones without dealing with common bile duct stones

ELIGIBILITY:
Inclusion Criteria:

* Patients with asymptomatic common bile duct stones.
* Patients with normal bilirubin levels.
* Patients with normal alkaline phosphates level.

Exclusion Criteria:

* Patients with history of jaundice.
* Patients with abnormal liver functions.

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: patients presented by chronic calcular cholecystitis and during investigation they discovers that they have silent common bile duct stones
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
number of patients developed jaundice post cholecystectomy | 6 months
  patients presented by symptomatic gall bladder stones and during investigation discovered that they have silent common bile duct stone so we assess the safety of performing cholecystectomy without developing jaundice

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qeft Teatching Hospital, Qina
  - Qena Faculty of Medicine, Qina
  - Suez Faculty of Medicine, Suez

REFERENCES:
- [Derived] Maklad AA, Eltantawy M, Siam M, Abdelshafy M. Feasibility of cholecystectomy in patients with silent common bile duct stones cohort prospective single arm multicentre study. BMC Gastroenterol. 2025 Mar 11;25(1):158. doi: 10.1186/s12876-024-03459-6. PMID 40069599